CLINICAL TRIAL: NCT04168424
Title: Validation of the English Version of the FIMA Questionnaire
Acronym: FIMAEN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 103/2019
Record Dates: First submitted 2019-11-11; First posted 2019-11-19 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Elderly Persons
Keywords: resource use; assessment; elderly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — Completing the questionnaire for health-related resource use in the elderly population (FIMA) by the elderly people

SUMMARY:
The purpose of this study was to determine the validity and reliability of the English version of the Questionnaire for Health-Related Resource Use in an Elderly Population (FIMA).

ELIGIBILITY:
Inclusion Criteria:

-65+.

Exclusion Criteria:

* younger than 65+
* severe visual impairment
* severe auditory impairment
* poor command of English
* no consent to participate in the study

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: 60 elderly people 65 years of age and older, who will be admitted within the previous 48 hours to Gessler Clinic USA, will be recruited. The participants will be excluded if they have severe visual or auditory impairment, are likely to pass away within 24 hours, have a poor command of English, or are unwilling to participate. No individuals with cognitive impairments will be included in this study. Each patient will be evaluated twice: once within 48 hours at admission and once after two weeks.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Good validity and reliability of the FIMA | 11.2019-12.2020
  The Questionnaire for Health-Related Resource Use in an Elderly Population is a self-administered questionnaire, which assesses nine features and contains 28 questions altogether: questions 1-18 refer directly to the use of medical and nonmedical services by the elderly, whereas questions 19-28 concern the sociodemographic characteristics of the person surveyed as well as an assessment of questionnaire difficulty and time spent completing it.
  A total of minimum 60 elderly people, 65 years of age and older, who will be admitted to the Gessler Clinic, USA California, are recruited. All patients will be screening twice for health-related resource use, using the English version of the Questionnaire for Health-Related Resource Use in an Elderly Population. Each patient will be evaluated twice: once within 48 hours at admission and once after two weeks.
  The English FIMA demonstrate very good test-retest reliability, good validity, and ease of use for elderly people.

CONTACTS AND LOCATIONS:
Locations (1):
- Gessler Clinic, Winter Haven, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mazurek J, Sutkowska E, Szczesniak D, Urbanska KM, Rymaszewska J. FIMA, the questionnaire for health-related resource use in the elderly population: validity, reliability, and usage of the Polish version in clinical practice. Clin Interv Aging. 2018 Apr 27;13:787-795. doi: 10.2147/CIA.S158951. eCollection 2018. PMID 29731618
- [Background] Seidl H, Hein L, Scholz S, Bowles D, Greiner W, Brettschneider C, Konig HH, Holle R. [Validation of the FIMA Questionnaire for Health-Related Resource Use Against Medical Claims Data: The Role Played by Length of Recall Period]. Gesundheitswesen. 2021 Jan;83(1):66-74. doi: 10.1055/a-1010-6315. Epub 2019 Nov 7. German. PMID 31698476